CLINICAL TRIAL: NCT00218907
Title: An Educational HIV Pre-Test Counseling Video Program for Off Hours Testing in the ED: A Randomized Control Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: North Bronx Healthcare Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 03-073
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: HIV Counseling and Testing; HIV Infections
Keywords: HIV prevention; HIV counseling; HIV testing; Emergency Medicine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Procedure: Educational video

SUMMARY:
This study compared the educational effectiveness of a ten-minute pre-test counseling video with the usual practice of a session with an HIV counselor.

DETAILED DESCRIPTION:
HIV is increasingly affecting urban populations, making the inner city ED a prime venue for C&T because of their unique opportunity to identify HIV positive patients. These underserved communities often use the ED for their regular health care specifically because it provides services outside of the usual weekday working hours. However, there are significant barriers to HIV C&T in the ED, such as the lack of resources to provide prevention oriented messages, cost issues, and the feasibility of providing the required manpower for testing. The objective of this study is to determine whether an educational video, with the required pre-test counseling elements, conveys the necessary information for inner city ED patients to consent to a standard Elisa HIV test.

In order to address the HIV testing needs of the patient population presenting to the ED, innovative methods must be developed to provide HIV C&T, while simultaneously removing the barriers to testing. Video technology may provide an opportunity to make HIV counseling feasible when counselors are not available.

ELIGIBILITY:
Inclusion Criteria:

* All patients awaiting UC treatment were approached for the study.
* Patients 18 years of age and older were included
* Patients who spoke English and Spanish were included.

Exclusion Criteria:

* Clinically unstable,
* Diagnosed with HIV
* Unable to understand the consent process because such patients require unique arrangements for consenting processes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2003-06; Study Completion 2003-08

PRIMARY OUTCOMES:
Comparison of mean knowledge score in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD, MS, Principal Investigator — Jacobi Medical Center, Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States